CLINICAL TRIAL: NCT02981225
Title: Descriptive Study of a Phytotherapy Management Strategy for Mild to Moderate Major Depression With Phytostandard® Rhodiola-Saffron : a Combination of Rhodiola and Saffron Extracts.
Brief Title: Management Strategy for Mild to Moderate Major Depression: Combination of Rhodiola and Saffron Extracts.
Status: Completed | Type: Observational
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Other Study IDs: PiL-Obs-RSDep-015
Record Dates: First submitted 2016-11-24; First posted 2016-12-05 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Mild to Moderate Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Phytostandard® Rhodiola-Saffron

SUMMARY:
The purpose of the study is to describe, over 6 weeks, the evolution of depressive symptoms in patients with mild to moderate major depression in a strategy with Phytostandard® Rhodiola-Saffron supplementation

DETAILED DESCRIPTION:
For this study, 52 patients are going to be included. They will have a supplementation of Phytostandard® rhodiola/saffron, from 2 tablets per day during 42 days.

on the one hand, during the two visits (inclusion and follow-up), the investigator completes the Hamilton Depression Scale (HAM-D) and the Clinical Global Impression (CGI). During the inclusion visit, he completes with his patient CIM-10 for depression diagnostic.

on the other hand, patients complete HAD 4 times : just after the inclusion visit, at day 14, at day 28 and just before the follow-up visit. He completes the Patient Global Impression too at each time.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from mild to moderate depression as defined in CIM-10
* Having a score on the HAM-D questionnaire between 8 and 18
* Having agreed to participate at the study after being informed by the investigator

Exclusion Criteria:

* Depressive patients already under medication or discontinuation of medication less than a month ago
* Patients with severe depression as defined in CIM-10 or HAM-D> 18
* Patients considered at risk: attempted suicide or suicidal (observed by the investigator or Hamilton item 3 score> 2)
* Patients with psychiatric disorders: schizophrenia, bipolarity, addiction (drugs, alcohol ...), etc.
* Patient with severe disease (cancer, kidney or heart disease) or patient with a contra-indication for taking the product (patient under anti-hypertensive ...)
* Patients using agents containing piperine or St. John's wort (interactions)
* Pregnant or breastfeeding patients
* Patients who do not wish to complement Phytostandard® Rhodiola - Saffron.
* Patients who do not wish to participate in the study.
* Patients unable to understand the ins and outs of the study (mental incapacity, language barrier).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from mild to moderate depression
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Evolution of HAM-D scale | between day 0 and day 42

SECONDARY OUTCOMES:
Evolution of HAD patient scale | between day 0 and day 42
Evolution of CGI | between day 0 and day 42
Evolution of PGI | between day 0 and day 42

CONTACTS AND LOCATIONS:
Locations (1):
- Pileje, Paris, France